CLINICAL TRIAL: NCT04268056
Title: Characterization of Skin Microbiome Profile Before and During Radiation Therapy and it's Correlation to the Occurrence and Severity of Radiation Dermatitis
Brief Title: Characterization of Skin Microbiome Profile and it's Correlation to Radiation Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AceTech (Industry)
Responsible Party: Sponsor
Other Study IDs: 0141-19-RMB
Record Dates: First submitted 2020-02-06; First posted 2020-02-13 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Radiation Dermatitis
Keywords: Radiation dermatitis; Radio Therapy; Microbiome Profile
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Skin microbiome samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RT patients: 100 patients with breast cancer undergoing radiation therapy
  Interventions: Diagnostic Test: Collection of skin culture samples

INTERVENTIONS:
Diagnostic Test: Collection of skin culture samples — Collection of skin culture samples using a sterile swab. the swab will gently rubbed on the skin on the 3 different skin areas. The target areas are i) regions surrounding the RT treatment area (if possible, not from the scar area or from skin folds areas), ii) a control site of the normal (healthy) breast , iii) a control area on the forehead.

SUMMARY:
The purpose of this study is to characterize the skin microbiome profile of breast cancer patients before and after receiving Radio Therapy treatments, and evaluate the relationship between the microbiome profile and radiation dermatitis severity (grade) that the patient will develop. Such characterizations can lead to potential biomarkers and/or therapeutic targets that can be used for the prognosis, prevention and treatment of this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histological confirmation of breast malignancy
3. Primary or recurrent disease eligible
4. Patients after breast lumpectomy and that scheduled to receive radiotherapy
5. Patients that receive minimum of 45 Gy
6. Ability to complete questionnaire(s) by themselves or with assistance
7. Provide informed written consent

Exclusion Criteria:

1. Patients with prior radiotherapy to any portion of the planned treatment site
2. Tumour involvement of the skin
3. Patients with active rash, pre-existing dermatitis, lupus, or scleroderma
4. Patient with other skin diseases/ skin disorders
5. Recent use of systemic or topical antibiotics or antifungal medications within 21 days of first swab collection.
6. Recent use of any of the following within 21 days of first swab collection: o Systemic or topical steroids o Use of systemic immunosuppressant drugs o Use of ultraviolet light therapy
7. Prior usage of other topical and systemic medications within 21 days of first swab collection
8. Prior usage of topical cosmetic products, creams, lotions, or gels within 14 days of first swab collection in areas where samples are taken.
9. Clinical evidence of infection that in the judgement of the principle investigator would interfere with proper assessment of the skin microbiome
10. Prior organ or bone marrow transplant
11. Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the patient safety

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer undergoing radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Radiation Dermatitis grade | through study completion, an average of 1 year
  Study participant will be evaluated by physician and nurse for the occurrence and the severity of RD. Skin condition (grade of RD) in the radiation area will be measured by the Radiation Therapy Oncology Group (RTOG) scoring.
Microbiome composition | through study completion, an average of 1 year
  Collection of skin culture samples from body regions surrounding the RT treatment area and a control area

SECONDARY OUTCOMES:
Validation Procedure of evaluation of Radiation Dermatitis grade by the our application (Radia-App) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roxolyana Abdah-Borthnyak, MD, Principal Investigator — Director, Radiation Service for Female Cancer
Locations (1):
- Rambam Medical Center, Haifa, Israel